CLINICAL TRIAL: NCT01010126
Title: A Phase 2 Trial of Temsirolimus and Bevacizumab in Patients With Endometrial, Ovarian, Hepatocellular Carcinoma, Carcinoid or Islet Cell Cancer
Brief Title: Temsirolimus and Bevacizumab in Treating Patients With Advanced Endometrial, Ovarian, Liver, Carcinoid, or Islet Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02086; NCI-2012-02086 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-2011-02504; MC0845; CDR0000653790; NCI-2012-01049; 8233 (Other: Mayo Clinic); 8233 (Other: CTEP); N01CM00032 (NIH); N01CM00038 (NIH); N01CM00039 (NIH); N01CM00070 (NIH); N01CM00071 (NIH); N01CM00099 (NIH); N01CM00100 (NIH); N01CM62201 (NIH); N01CM62203 (NIH); N01CM62204 (NIH); N01CM62205 (NIH); N01CM62206 (NIH); N01CM62207 (NIH); N01CM62208 (NIH); N01CM62209 (NIH); P30CA015083 (NIH); P50CA102701 (NIH)
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Results first posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Adult Hepatocellular Carcinoma; Advanced Adult Hepatocellular Carcinoma; Endometrial Serous Adenocarcinoma; Localized Non-Resectable Adult Liver Carcinoma; Lung Carcinoid Tumor; Malignant Pancreatic Gastrinoma; Malignant Pancreatic Glucagonoma; Malignant Pancreatic Insulinoma; Malignant Pancreatic Somatostatinoma; Metastatic Digestive System Neuroendocrine Tumor G1; Ovarian Carcinosarcoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Seromucinous Carcinoma; Ovarian Serous Surface Papillary Adenocarcinoma; Pancreatic Alpha Cell Adenoma; Pancreatic Beta Cell Adenoma; Pancreatic Delta Cell Adenoma; Pancreatic G-Cell Adenoma; Pancreatic Polypeptide Tumor; Recurrent Adult Liver Carcinoma; Recurrent Digestive System Neuroendocrine Tumor G1; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Pancreatic Neuroendocrine Carcinoma; Recurrent Primary Peritoneal Carcinoma; Recurrent Uterine Corpus Carcinoma; Regional Digestive System Neuroendocrine Tumor G1; Stage IIIA Fallopian Tube Cancer; Stage IIIA Ovarian Cancer; Stage IIIA Primary Peritoneal Cancer; Stage IIIA Uterine Corpus Cancer; Stage IIIB Fallopian Tube Cancer; Stage IIIB Ovarian Cancer; Stage IIIB Primary Peritoneal Cancer; Stage IIIB Uterine Corpus Cancer; Stage IIIC Fallopian Tube Cancer; Stage IIIC Ovarian Cancer; Stage IIIC Primary Peritoneal Cancer; Stage IIIC Uterine Corpus Cancer; Stage IV Fallopian Tube Cancer; Stage IV Ovarian Cancer; Stage IV Primary Peritoneal Cancer; Stage IVA Uterine Corpus Cancer; Stage IVB Uterine Corpus Cancer; Uterine Carcinosarcoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Fallopian Tube Neoplasms; Ovarian Neoplasms; Somatostatinoma | interventions — Bevacizumab; Immunoglobulin G; Disulfides; temsirolimus; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (temsirolimus, bevacizumab) (Experimental): Patients receive temsirolimus IV on days 1, 8, 15, and 22, and bevacizumab IV over 30-90 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Temsirolimus

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar FKB238; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
Drug: Temsirolimus — Given IV
  Other Names: CCI-779; CCI-779 Rapamycin Analog; Cell Cycle Inhibitor 779; Rapamycin Analog; Rapamycin Analog CCI-779; Torisel

SUMMARY:
This phase II trial studies how well temsirolimus and bevacizumab work in treating patients with advanced endometrial, ovarian, liver, carcinoid, or islet cell cancer. Temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of cancer by blocking blood flow to the tumor. Giving temsirolimus together with bevacizumab may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the response rate and progression-free survival at 6 months in patients with endometrial, ovarian, hepatocellular carcinoma, carcinoid or islet cell cancer.

II. To determine the toxicity of the combination of temsirolimus and bevacizumab in patients with endometrial, ovarian, hepatocellular carcinoma, carcinoid or islet cell cancer.

SECONDARY OBJECTIVES:

I. To collect blood and tumor specimens from all patients entered on the trial for possible future analysis.

OUTLINE:

Patients receive temsirolimus intravenously (IV) on days 1, 8, 15, and 22, and bevacizumab IV over 30-90 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed endometrial (endometrioid, uterine, papillary serous carcinoma, and carcinosarcoma), ovarian (primary peritoneal/fallopian tube, serous, endometrioid, mixed, and poorly differentiated epithelial ovarian cancers [for purposes of eligibility, carcinosarcoma is considered a poorly differentiated carcinoma]), hepatocellular carcinoma, carcinoid or islet cell (neuroendocrine: well- or moderately-differentiated neuroendocrine) cancer which are locally advanced, recurrent, or metastatic
* Patients must have measurable disease; patients having only lesions measuring >= 1 cm to < 2 cm must use spiral computed tomography (CT) imaging for both pre- and post-treatment tumor assessments; patients who have had prior palliative radiotherapy to metastatic lesion(s) must have at least one measurable lesion(s) that have not been previously irradiated
* Radiation therapy (adjuvant or palliative) must be completed >= 4 weeks prior to registration, if applicable
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelets >= 75,000/mm^3
* Hemoglobin >= 9.0 g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN); Note: direct bilirubin and international normalized ratio (INR) for hepatocellular carcinoma (HCC) patients allowed as per Child-Turcotte-Pugh scoring
* Alkaline phosphatase =< 2.5 x ULN (=< 5 x ULN if liver metastasis is present or patient is in HCC cohort)
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 2.5 x ULN (=< 5 x ULN if liver metastasis is present or patient is in HCC cohort)
* Creatinine =<1.5 x ULN
* Urinalysis < 2+ protein; urine protein should be screened by dipstick or urine analysis; for proteinuria >= 2+, 24-hour urine protein should be obtained and the level should be < 2 g for patient enrollment
* Fasting serum cholesterol =< 350 mg/dL (=< 9.0 mmol/L)
* Triglycerides =< 1.5 x ULN (mg/dL or mmol/L); patients with triglyceride levels > 1.5 x ULN can be started on lipid lowering agents and reevaluated within 1 week; if levels go to =< 1.5 x ULN, they can be considered for the trial and continue the lipid lowering agents; NOTE: cholesterol and triglyceride measurement and management are not required for single-agent bevacizumab cohort with islet cell carcinoma
* International normalized ratio (INR) =< 1.5 (unless the patient is on full dose warfarin)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1
* Capable of understanding the investigational nature, potential risks and benefits of the study and able to provide valid informed consent
* Negative serum pregnancy test done =< 7 days prior to registration, for women of childbearing potential only; NOTE: patients and their partners should be practicing an effective form of contraception during the study and for at least 3 months following the last dose of this combined therapy
* Full-dose anticoagulants, if a patient is receiving full-dose anticoagulants (except carcinoid tumors), the following criteria should be met for enrollment: the subject must have an in-range INR (usually between 2 and 3) on a stable dose of warfarin or on stable dose of low molecular weight (LMW) heparin
* Prior systemic treatments for metastatic disease are permitted, including targeted therapies, biologic response modifiers, chemotherapy, hormonal therapy, or investigational therapy; exception: in the case of endometrial cancer no prior chemotherapy for metastatic or recurrent disease is allowed; prior planned adjuvant chemotherapy is allowed
* Patients who have had prior anthracycline must have a normal ejection fraction on left ventricular ejection fraction (LVEF) assessment by multigated acquisition scan (MUGA) or echocardiogram (Echo) =< 4 weeks prior to registration
* Availability of tissue if applicable (from the primary tumor or metastases) for tumor studies for banking; Note: in the case of hepatocellular cancer if diagnosed by clinical and radiologic criteria only, availability of tissue not applicable
* Willingness to donate blood for biomarker studies related to the type of therapies used in this trial and the tumor types being treated
* ENDOMETRIAL CANCER (PERMANENTLY CLOSED TO ENROLLMENT)
* Any hormonal therapy directed at the malignant tumor is allowed; NOTE: therapy must be discontinued at least one week prior to registration
* Prior systemic therapy including biologic and immunologic agents as adjuvant treatment, must be discontinued at least 3 weeks prior to registration
* Recurrent or persistent endometrial adenocarcinoma, uterine papillary serous carcinoma and carcinosarcoma which is refractory to curative therapy or established treatments; NOTE: histologic or cytologic confirmation of original primary tumor is required
* HEPATOCELLULAR CANCER (PERMANENTLY CLOSED TO ENROLLMENT)
* HCC confirmed by biopsy OR diagnosed by clinical and radiologic criteria; all of the following criteria must be met or a biopsy is required:

  * Known cirrhosis or chronic hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
  * Hypervascular liver masses > 2 cm, and either serum alpha-fetoprotein (AFP) > 400 ng/ml, or
  * AFP > three times normal and doubling in value in the antecedent 3 months
* Child-Pugh A (=< 6 points) or better liver status
* Prior regional treatments for liver metastasis are permitted including:

  * Selective internal radiation therapy such as brachytherapy, cyberknife, radiolabeled microsphere embolization, etc.
  * Hepatic artery chemoembolization
  * Hepatic artery embolization
  * Hepatic artery infusional chemotherapy
  * Radiofrequency ablation NOTE: patients must be >= 4 weeks from treatment and show progressive disease in the liver after regional therapy or must have measurable disease outside the liver
* Concomitant anti-viral therapy is allowed
* History of prior varices or evidence of varices on pre-study CT/magnetic resonance imaging (MRI) imaging are required to undergo endoscopy =< 4 weeks prior to registration; those who had received specific therapy (banding and/or sclerotherapy) and had not bled within the prior 6 months are eligible
* Suitably recovered from prior localized therapy, in the opinion of the investigator
* ISLET CELL CANCER AND CARCINOID TUMOR (PERMANENTLY CLOSED TO ENROLLMENT)
* Patient has evidence of progressive disease as documented by Response Evaluation Criteria in Solid Tumors (RECIST) =< 7 months prior to study entry
* Carcinoid tumor cohort: prior and concurrent long-acting somatostatin analogue therapy is required; patient has to be on a stable dose of a long-acting somatostatin analogue >= 2 months prior to study entry with documentation of progressive disease on current dose
* Islet cell tumor cohort: prior and/or concurrent long-acting somatostatin analogue therapy is allowed, but not required; if patient is continued on a long-acting somatostatin analogue, a stable dose for >= 2 months prior to study entry is required with documentation of progressive disease on current dose
* Prior therapies allowed include:

  * =< 2 prior chemotherapy regimens
  * Prior interferon >= 4 weeks prior to registration
  * Radiolabeled octreotide therapy (patients with prior radiolabeled octreotide therapy should have progressive disease after such therapy)
  * Other investigational therapy NOTE: islet Cell Single Agent Bevacizumab Cohort: Prior mammalian target of rapamycin (mTOR) inhibitor is allowed
* Prior regional treatments for liver metastasis are permitted including:

  * Selective internal radiation therapy such as brachytherapy, cyberknife, radiolabeled microsphere embolization, etc.
  * Hepatic artery chemoembolization
  * Hepatic artery embolization
  * Hepatic artery infusional chemotherapy
  * Radiofrequency ablation NOTE: patients must be >= 12 weeks from treatment and show progressive disease in the liver after regional therapy or must have measurable disease outside the liver

Exclusion Criteria:

* Prior therapy with vascular endothelial growth factor receptor (VEGFR) targeting agents or mammalian target of rapamycin (mTOR) inhibitors (except as in HCC and in the Islet cell single agent bevacizumab alone cohort where prior mTOR inhibitor is allowed); Note: prior use of bevacizumab is not allowed in any cohort
* Invasive procedures defined as follows:

  * Major surgical procedure, open biopsy or significant traumatic injury =< 4 weeks prior to registration
  * Anticipation of need for major surgical procedures during the course of the study
  * Core biopsy =< 7 days prior to registration
* Serious or non-healing wound, ulcer or bone fracture
* History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess =< 180 days prior to first date of bevacizumab therapy
* Evidence of bleeding diathesis or coagulopathy in the absence of therapeutic anticoagulation
* Evidence of a history bleeding =< 6 months such as hemoptysis, or cerebrovascular accident =< previous 6 months, or peripheral vascular disease with claudication on < 1 block, or history of clinically significant bleeding, because of the potential bleeding and/or clotting risk with bevacizumab
* Untreated central nervous system (CNS) metastases; exceptions: patients with known CNS metastases can be enrolled if the brain metastases have been adequately treated and there is no evidence of progression or hemorrhage after treatment as ascertained by clinical examination and brain imaging (MRI or CT) =< 12 weeks prior to registration and no ongoing requirement for steroids

  * Anticonvulsants (stable dose) are allowed
  * Patients who had surgical resection of CNS metastases or brain biopsy =< 3 months prior to registration will be excluded
* Significant cardiovascular disease defined as congestive heart failure (New York Heart Association class II, III or IV), angina pectoris requiring nitrate therapy, or recent myocardial infarction (=< 6 months prior to registration)
* Uncontrolled hypertension (defined as a blood pressure of >= 150 mmHg systolic and/or >= 90 mmHg diastolic)
* Patient is on angiotensin-converting-enzyme (ACE) inhibitors (benazapril, captopril, enalopril, fosonopril, lisinopril, moexipril, perindopril, quinopril, ramipril, and trandolapril); (patients may have an alternate antihypertensive substituted); NOTE: ACE inhibitors are allowed in single agent bevacizumab cohort
* Currently active, second malignancy other than non-melanoma skin cancers; NOTE: patients are not considered to have a 'currently active' malignancy if they have completed anti-cancer therapy and are considered by their physician to be at less than 30% risk of relapse
* Any of the following, as this regimen may be harmful to a developing fetus or nursing child:

  * Pregnant women
  * Breastfeeding women
  * Men or women of childbearing potential or their sexual partners who are unwilling to employ adequate contraception (diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.) NOTE: the effects of the agent(s) on the developing human fetus at the recommended therapeutic dose are unknown
* Known hypersensitivity to other recombinant human antibodies or Chinese hamster ovary cell products
* Other uncontrolled serious medical or psychiatric condition (e.g. cardiac arrhythmias, diabetes, etc.)
* Current therapy with a cytochrome P450 3A4 (CYP3A4) inhibitor or inducer; NOTE: these agents are allowed in the single-agent bevacizumab islet cell carcinoma cohort
* Active infection requiring antibiotics
* Active bleeding or pathological conditions that carry high risk of bleeding (e.g. tumor involving major vessels, known varices)
* Known human immunodeficiency virus (HIV)-positive
* ENDOMETRIAL CANCER (PERAMANENTLY CLOSED TO ENROLLMENT)
* Received prior radiotherapy to any portion of the abdominal cavity or pelvis OTHER THAN for the treatment of endometrial cancer
* Any chemotherapy for metastatic or recurrent cancer
* Radiation therapy to > 25% of marrow bearing areas
* HEPATOCELLULAR CANCER EXCLUSION (PERMANENTLY CLOSED TO ENROLLMENT)
* Child-Pugh B or C classification
* Grade >= 3 hemorrhage =< 4 weeks prior to registration
* Prior liver transplant with evidence of recurrent or metastatic disease
* Patients on an active liver transplant list and considered likely to receive a liver transplant =< 6 months following registration
* Clinical evidence of encephalopathy
* Prior treatment with sorafenib or other vascular endothelial growth factor (VEGF) inhibitors; NOTE: Exceptions allowed for patients unable to tolerate the agent; intolerance is defined in this protocol as a discontinued agent due to side effects with an exposure < to 4 weeks of drug, at any dose level
* OVARIAN CANCER (PERMANENTLY CLOSED TO ENROLLMENT)
* Clinical signs and symptoms of gastrointestinal (GI) obstruction and require parental hydration/nutrition or tube feeding
* Evidence of free abdominal air not explained by paracentesis or recent surgical procedures
* Received more than two prior cytotoxic chemotherapy regimens for persistent or recurrent disease
* CARCINOID (PERMANENTLY CLOSED TO ENROLLMENT)
* Patients on anticoagulant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2009-09-08; Primary Completion 2017-03-13 (Actual); Study Completion 2017-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Pitot, Principal Investigator — Mayo Clinic
Locations (61):
- United States (57):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Tower Cancer Research Foundation, Beverly Hills, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - City of Hope South Pasadena, South Pasadena, California
  - University of Connecticut, Farmington, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Maryland Saint Joseph Medical Center, Towson, Maryland
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Memorial Sloan Kettering Sleepy Hollow, Sleepy Hollow, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
- Canada (4):
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Trillium Health Partners - Credit Valley Hospital, Mississauga, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Abuzakhm SM, Sukrithan V, Fruth B, Qin R, Strosberg J, Hobday TJ, Semrad T, Reidy-Lagunes D, Kindler HL, Kim GP, Knox JJ, Kaubisch A, Villalona-Calero M, Chen H, Erlichman C, Shah MH. A phase II study of bevacizumab and temsirolimus in advanced extra-pancreatic neuroendocrine tumors. Endocr Relat Cancer. 2023 Sep 13;30(11):e220301. doi: 10.1530/ERC-22-0301. Print 2023 Nov 1. PMID 37702588
- [Derived] Hobday TJ, Qin R, Reidy-Lagunes D, Moore MJ, Strosberg J, Kaubisch A, Shah M, Kindler HL, Lenz HJ, Chen H, Erlichman C. Multicenter Phase II Trial of Temsirolimus and Bevacizumab in Pancreatic Neuroendocrine Tumors. J Clin Oncol. 2015 May 10;33(14):1551-6. doi: 10.1200/JCO.2014.56.2082. Epub 2014 Dec 8. PMID 25488966
- [Derived] Knox JJ, Qin R, Strosberg JR, Tan B, Kaubisch A, El-Khoueiry AB, Bekaii-Saab TS, Rousey SR, Chen HX, Erlichman C. A phase II trial of bevacizumab plus temsirolimus in patients with advanced hepatocellular carcinoma. Invest New Drugs. 2015 Feb;33(1):241-6. doi: 10.1007/s10637-014-0169-3. Epub 2014 Oct 16. PMID 25318437

RESULTS

PARTICIPANT FLOW:
Groups:
- Endometrial Cohort; Ovarian Cohort; Hepatocellular Cohort; Carcinoid Cohort; Islet Cell (Double Agent) Cohort: Patients receive 25 mg temsirolimus IV on days 1, 8, 15, and 22, and 10 mg/kg bevacizumab IV over 30-90 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Islet Cell (Bevacizumab-only) Cohort: Patients receive 10 mg/kg bevacizumab IV over 30-90 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Endometrial Cohort | Ovarian Cohort | Hepatocellular Cohort | Carcinoid Cohort | Islet Cell (Double Agent) Cohort | Islet Cell (Bevacizumab-only) Cohort
Started | 27 | 58 | 28 | 57 | 58 | 24
Completed | 26 | 58 | 27 | 57 | 55 | 24
Not Completed | 1 | 0 | 1 | 0 | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Endometrial Cohort | Ovarian Cohort | Hepatocellular Cohort | Carcinoid Cohort | Islet Cell (Double Agent) Cohort | Islet Cell (Bevacizumab-only) Cohort | Total
Number analyzed (Participants) | 26 | 58 | 27 | 57 | 58 | 24 | 250
Age, Continuous [Median (Full Range); unit: years] | 60 [40 to 80] | 62.5 [35 to 82] | 59 [31 to 74] | 62 [35 to 89] | 58.5 [29 to 81] | 54.5 [40 to 78] | 60 [29 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 58 | 5 | 31 | 29 | 10 | 159
  Male | 0 | 0 | 22 | 26 | 29 | 14 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 2 | 0 | 1 | 2 | 11
  Not Hispanic or Latino | 19 | 54 | 25 | 54 | 57 | 22 | 231
  Unknown or Not Reported | 3 | 2 | 0 | 3 | 0 | 0 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 5 | 3 | 0 | 0 | 0 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 3 | 2 | 2 | 6 | 8 | 3 | 24
  White | 22 | 49 | 22 | 49 | 50 | 20 | 212
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 0 | 1 | 0 | 1 | 5
Region of Enrollment [Number; unit: participants]
  Canada | 5 | 34 | 8 | 2 | 14 | 0 | 63
  United States | 21 | 24 | 19 | 55 | 44 | 24 | 187

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival Rate
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. The 6-month progression free survival rate is the proportion of evaluable patients progression-free 6 months from registration. The 6-month progression-free rate is defined as the total number of efficacy evaluable patients on study without documentation of disease progression 6 months from registration divided by the total number of evaluable patients enrolled on study. Kaplan-Meier methodology will be used to estimate the final success proportion (i.e. progression free at 6 months with a 95% confidence interval).
Time Frame: 6 months
Population: All patients that received study treatment and were evaluated for response are included in this analysis
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Endometrial Cohort | Ovarian Cohort | Hepatocellular Cohort | Carcinoid Cohort | Islet Cell (Double Agent) Cohort | Islet Cell (Bevacizumab-only) Cohort
Number analyzed (Participants) | 26 | 58 | 27 | 55 | 54 | 24
proportion of patients | 0.52 [0.35 to 0.77] | 0.40 [0.29 to 0.55] | 0.71 [0.54 to 0.94] | 0.84 [0.75 to 0.95] | 0.85 [0.75 to 0.95] | 0.87 [0.74 to 1.00]

2. Primary Outcome: Tumor Response Rate
Description: Tumor response rate defined as the total number of efficacy-evaluable patients who achieved a complete or partial response according to the RECIST criteria divided by the total number of efficacy evaluable patients enrolled on study. Patients were evaluated using the Response Evaluation Criteria In Solid Tumors (RECIST) v1.1. In brief, a Complete Response (CR) means the complete disappearance of all target lesions and a reduction in each lymph node to <1 cm. A Partial Response (PR) is defined as a 30% decrease in the sum of the longest diameter of the non-nodal target lesion from baseline. Each requires no new lesions present at evaluation. The proportion of participants with a response is provided here for each cohort. The proportion was calculated as the number of patients that had a best response of CR or PR divided by the number of patients evaluated for a response in each cohort.
Time Frame: Up to 3 years
Population: For this analysis, the number of patients that had a best response of CR or PR were divided by the number of patients evaluated for a response.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Endometrial Cohort | Ovarian Cohort | Hepatocellular Cohort | Carcinoid Cohort | Islet Cell (Double Agent) Cohort | Islet Cell (Bevacizumab-only) Cohort
Number analyzed (Participants) | 26 | 58 | 27 | 57 | 58 | 24
proportion of participants | 0.31 [0.14 to 0.52] | 0.31 [0.20 to 0.45] | 0.19 [0.06 to 0.38] | 0.12 [0.05 to 0.24] | 0.40 [0.27 to 0.53] | 0.17 [0.05 to 0.37]

3. Secondary Outcome: Duration of Response
Description: Duration of response is defined for all evaluable patients who have achieved a response as the date at which the patient's objective status is first noted to be either a CR or PR to the date progression is documented. Objective response was assessed using Response Evaluation Criteria In Solid Tumors (RECIST) as described in Primary Objective 2 in this report. Median duration of response and the confidence interval for the median duration will be computed.
Time Frame: Time from date at which the patient's objective status is first noted to be either a complete response (CR) or partial response (PR) to the date progression is documented, assessed up to 3 years
Population: All patients that were assessed as a Complete Response or Partial Response were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Endometrial Cohort | Ovarian Cohort | Hepatocellular Cohort | Carcinoid Cohort | Islet Cell (Double Agent) Cohort | Islet Cell (Bevacizumab-only) Cohort
Number analyzed (Participants) | 8 | 18 | 5 | 7 | 23 | 4
months | 25.1 [0 to 35.5] | 6.4 [3.7 to 10.8] | 6.4 [0 to 11.1] | 15.0 [0 to 18.8] | 11.3 [8.8 to 21.2] | 10.9 [3.7 to 34.1]

4. Secondary Outcome: Incidence of Adverse Events
Description: Adverse events are defined as events that are classified as either possibly, probably, or definitely related to study treatment, graded per National Cancer Institute Common Terminology Criteria for Adverse Events Version 3.0. The number of patients reporting grade 3 or higher adverse events at least possibly related to treatment are reported here. For a complete list of all reported adverse events, please see the adverse events section of this report.
Time Frame: Every cycle of treatment, up to 3 years
Population: All patients that received protocol treatment and were evaluated for adverse events are reported in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Endometrial Cohort | Ovarian Cohort | Hepatocellular Cohort | Carcinoid Cohort | Islet Cell (Double Agent) Cohort | Islet Cell (Bevacizumab-only) Cohort
Number analyzed (Participants) | 26 | 58 | 27 | 57 | 55 | 24
Participants
  Grade 3 Adverse Event | 17 | 32 | 24 | 32 | 36 | 13
  Grade 4 Adverse Event | 1 | 6 | 0 | 6 | 8 | 0
  Grade 5 Adverse Event | 1 | 0 | 1 | 2 | 0 | 0

5. Secondary Outcome: Overall Survival
Description: Survival time will be defined as the time from registration to death. Time to event distributions will be estimated using the Kaplan-Meier method.
Time Frame: Time from registration to death, assessed up to 3 years
Population: All patients that received study intervention and were followed for survival were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Endometrial Cohort | Ovarian Cohort | Hepatocellular Cohort | Carcinoid Cohort | Islet Cell (Double Agent) Cohort | Islet Cell (Bevacizumab-only) Cohort
Number analyzed (Participants) | 26 | 58 | 27 | 57 | 58 | 24
months | 11.5 [6.5 to NA] — Too few deaths occurred to estimate an upper 95% CI. | 16.3 [11.1 to 21.9] | 14.8 [9.7 to 18.1] | 32.7 [25.2 to 38.3] | 35.0 [14.6 to NA] — Too few deaths occurred to estimate an upper 95% CI. | NA [30.6 to NA] — Too few deaths occurred to estimate a median or an upper 95% CI.

6. Secondary Outcome: Time to Disease Progression
Description: Time to progression is defined as the time from registration to disease progression. Patients who died without documentation of progression will be considered to have progressed on the date of their death. If a patient starts treatment and fails to return for evaluation, that patient will be censored for progression of disease at day one post-registration.
Time Frame: Time from registration to disease progression, assessed up to 3 years
Population: All patients that began protocol treatment and were evaluated for response are included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Endometrial Cohort | Ovarian Cohort | Hepatocellular Cohort | Carcinoid Cohort | Islet Cell (Double Agent) Cohort | Islet Cell (Bevacizumab-only) Cohort
Number analyzed (Participants) | 26 | 58 | 27 | 55 | 54 | 24
months | 6.0 [2.5 to 9.8] | 5.6 [4.3 to 6.4] | 8.0 [5.8 to 10.9] | 15.2 [11.4 to 24.2] | 13.1 [11.2 to 16.6] | 18.0 [10.6 to 37.0]

7. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure is defined as the time from study entry to the date patients end treatment.Time to treatment failure will be evaluated using the method of Kaplan-Meier.
Time Frame: Time from study entry to the date patients end treatment, assessed up to 3 years
Population: All patients that began study treatment were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Endometrial Cohort | Ovarian Cohort | Hepatocellular Cohort | Carcinoid Cohort | Islet Cell (Double Agent) Cohort | Islet Cell (Bevacizumab-only) Cohort
Number analyzed (Participants) | 26 | 58 | 27 | 55 | 54 | 24
months | 3.8 [2.3 to 6.4] | 4.5 [2.7 to 5.6] | 6.5 [2.3 to 8.0] | 5.5 [4.4 to 8.1] | 11.3 [8.6 to 13.3] | 11.8 [5.8 to 18.0]

ADVERSE EVENTS:
Time Frame: Adverse events were collected at the end of each 28 day cycle for a maximum of 58 cycles.
Description: Adverse events were collected at the end of each 28 day cycle for a maximum of 58 cycles.
Arm/Group | Endometrial Cohort | Ovarian Cohort | Hepatocellular Cohort | Carcinoid Cohort | Islet Cell (Double Agent) Cohort | Islet Cell (Bevacizumab-only) Cohort
All-Cause Mortality (participants affected / at risk) | 2/26 | 1/58 | 3/27 | 3/57 | 0/55 | 0/24
Serious Adverse Events (participants affected / at risk) | 16/26 | 34/58 | 13/27 | 36/57 | 27/55 | 6/24
Other Adverse Events (participants affected / at risk) | 26/26 | 58/58 | 27/27 | 56/57 | 55/55 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endometrial Cohort (N=26) | Ovarian Cohort (N=58) | Hepatocellular Cohort (N=27) | Carcinoid Cohort (N=57) | Islet Cell (Double Agent) Cohort (N=55) | Islet Cell (Bevacizumab-only) Cohort (N=24)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (5) | 2 (3) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Cardiac pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 5 (7) | 3 (3) | 8 (10) | 6 (6) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Esophageal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Esophageal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 2 (2) | 3 (4) | 2 (2) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 4 (5) | 0 (0) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (5) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Disease progression (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 4 (4) | 3 (4) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Ill-defined disorder (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sudden death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visceral edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic hemorrhage (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorectal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gallbladder infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bilirubin increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Laboratory test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Leukocyte count decreased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serum cholesterol increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight gain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 1 (2) | 5 (6) | 1 (1) | 0 (0)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Serum glucose decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (1) | 2 (3) | 3 (3) | 0 (0)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (5) | 2 (3) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Protein urine positive (Renal and urinary disorders) | 2 (3) | 2 (4) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urogenital disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal fistula (Reproductive system and breast disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Visceral arterial ischemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endometrial Cohort (N=26) | Ovarian Cohort (N=58) | Hepatocellular Cohort (N=27) | Carcinoid Cohort (N=57) | Islet Cell (Double Agent) Cohort (N=55) | Islet Cell (Bevacizumab-only) Cohort (N=24)
Blood disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 20 (79) | 48 (212) | 23 (122) | 49 (382) | 49 (556) | 8 (82)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (9) | 1 (10) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Lymphatic disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (13) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 1 (7) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac pain (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (3) | 0 (0)
Hearing loss (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Hearing test abnormal (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (8) | 0 (0) | 1 (1) | 1 (7) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry eye syndrome (Eye disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye disorder (Eye disorders) | 1 (45) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flashing vision (Eye disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 3 (8) | 0 (0) | 2 (8) | 2 (2) | 0 (0)
Watering eyes (Eye disorders) | 4 (13) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 3 (5) | 0 (0) | 3 (9) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 13 (21) | 4 (8) | 11 (27) | 7 (19) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (3) | 0 (0) | 0 (0)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Anal mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal pain (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 1 (5) | 1 (1)
Anal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 7 (25) | 11 (16) | 3 (5) | 7 (10) | 9 (17) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 9 (36) | 18 (39) | 7 (20) | 33 (113) | 21 (73) | 5 (20)
Dry mouth (Gastrointestinal disorders) | 4 (10) | 4 (28) | 1 (3) | 5 (24) | 1 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (5) | 5 (6) | 2 (6) | 4 (12) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (6) | 2 (5) | 0 (0) | 1 (1) | 3 (15) | 0 (0)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 12 (31) | 18 (44) | 4 (6) | 28 (76) | 33 (116) | 3 (23)
Esophageal mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 3 (7) | 2 (2) | 0 (0)
Gastric mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (3) | 3 (6) | 1 (1) | 7 (7) | 5 (8) | 2 (2)
Gastroscopy abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 3 (15) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 10 (15) | 4 (8) | 0 (0)
Lip pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (9) | 2 (3) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 5 (13) | 27 (86) | 11 (27) | 17 (25) | 12 (43) | 2 (2)
Nausea (Gastrointestinal disorders) | 11 (63) | 24 (49) | 9 (22) | 23 (63) | 22 (69) | 4 (13)
Oesophagoscopy abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 1 (2) | 3 (10) | 1 (1) | 1 (1) | 2 (8) | 0 (0)
Oral pain (Gastrointestinal disorders) | 5 (6) | 5 (6) | 2 (4) | 7 (17) | 3 (13) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (3) | 4 (4) | 1 (2) | 5 (10) | 2 (3) | 0 (0)
Rectal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (4) | 2 (2) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 2 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 3 (3) | 2 (2) | 4 (8) | 5 (12) | 8 (21) | 0 (0)
Vomiting (Gastrointestinal disorders) | 7 (10) | 8 (13) | 5 (8) | 13 (24) | 17 (26) | 3 (5)
Chest pain (General disorders) | 1 (2) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 0 (0)
Chills (General disorders) | 3 (4) | 5 (12) | 0 (0) | 4 (7) | 2 (2) | 0 (0)
Edema limbs (General disorders) | 5 (22) | 8 (25) | 3 (8) | 12 (55) | 15 (70) | 2 (2)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 21 (120) | 43 (152) | 14 (67) | 40 (236) | 48 (293) | 12 (70)
Fever (General disorders) | 0 (0) | 4 (4) | 3 (4) | 5 (6) | 4 (4) | 1 (1)
Flu-like symptoms (General disorders) | 2 (2) | 1 (3) | 0 (0) | 1 (1) | 1 (3) | 1 (1)
Gait abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
General symptom (General disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (8) | 2 (15) | 0 (0)
Ill-defined disorder (General disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 2 (7) | 1 (1) | 2 (4) | 2 (3) | 0 (0)
Pain (General disorders) | 4 (5) | 3 (7) | 1 (1) | 3 (31) | 11 (57) | 2 (2)
Hypersensitivity (Immune system disorders) | 0 (0) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Immune system disorder (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1) | 4 (6) | 3 (3) | 3 (6) | 3 (3)
Joint infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nail infection (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (6) | 1 (1)
Skin infection (Infections and infestations) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (5) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (4) | 1 (1) | 2 (5) | 2 (3) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (2) | 5 (9) | 0 (0) | 3 (9) | 4 (18) | 1 (2)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Tracheal hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 2 (8) | 2 (4) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2) | 1 (1) | 0 (0) | 4 (6) | 3 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 9 (28) | 14 (24) | 6 (33) | 18 (62) | 25 (113) | 3 (6)
Alkaline phosphatase increased (Investigations) | 7 (33) | 13 (24) | 3 (17) | 20 (114) | 19 (76) | 3 (22)
Aspartate aminotransferase increased (Investigations) | 11 (40) | 20 (43) | 8 (47) | 24 (100) | 31 (120) | 4 (9)
Bilirubin increased (Investigations) | 1 (2) | 2 (2) | 9 (21) | 14 (48) | 14 (40) | 1 (1)
Creatinine increased (Investigations) | 4 (20) | 9 (29) | 2 (7) | 18 (60) | 9 (42) | 4 (7)
Fibrinogen decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
INR increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (8) | 1 (1) | 0 (0)
Laboratory test abnormal (Investigations) | 1 (1) | 1 (2) | 0 (0) | 4 (7) | 2 (2) | 0 (0)
Leukocyte count decreased (Investigations) | 10 (26) | 30 (108) | 16 (91) | 38 (158) | 34 (289) | 3 (12)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 6 (14) | 7 (11) | 6 (21) | 16 (72) | 19 (99) | 0 (0)
Neutrophil count decreased (Investigations) | 10 (15) | 25 (55) | 15 (54) | 21 (62) | 28 (130) | 3 (5)
Platelet count decreased (Investigations) | 16 (53) | 27 (86) | 22 (159) | 50 (327) | 41 (479) | 7 (52)
Serum cholesterol increased (Investigations) | 22 (147) | 38 (162) | 12 (49) | 38 (231) | 46 (408) | 7 (10)
Weight gain (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Weight loss (Investigations) | 8 (15) | 9 (29) | 6 (30) | 20 (73) | 12 (38) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 16 (39) | 23 (59) | 8 (28) | 27 (72) | 29 (70) | 5 (14)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 10 (43) | 14 (24) | 4 (7) | 30 (159) | 28 (138) | 11 (33)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (3) | 7 (8) | 0 (0)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Serum albumin decreased (Metabolism and nutrition disorders) | 3 (15) | 6 (7) | 3 (11) | 13 (37) | 13 (49) | 2 (2)
Serum calcium decreased (Metabolism and nutrition disorders) | 3 (4) | 5 (10) | 2 (2) | 10 (23) | 11 (61) | 1 (1)
Serum calcium increased (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 6 (10)
Serum glucose decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 1 (3) | 6 (8) | 1 (2) | 4 (9) | 1 (4) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 2 (3) | 4 (4) | 3 (3) | 10 (25) | 10 (22) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 7 (10) | 10 (15) | 2 (2) | 25 (63) | 11 (25) | 3 (4)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3) | 4 (4) | 2 (2) | 5 (5)
Serum sodium decreased (Metabolism and nutrition disorders) | 2 (2) | 5 (8) | 3 (4) | 6 (15) | 14 (42) | 5 (5)
Serum sodium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Serum triglycerides increased (Metabolism and nutrition disorders) | 16 (115) | 25 (73) | 7 (18) | 29 (176) | 32 (172) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (12) | 5 (5) | 5 (5) | 3 (5) | 3 (3) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Joint disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 5 (41) | 5 (7) | 2 (7) | 3 (4) | 3 (11) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (7) | 0 (0) | 4 (4) | 3 (4) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 1 (3) | 2 (2) | 0 (0) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 6 (11) | 6 (16) | 4 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (16) | 6 (9) | 0 (0) | 1 (5) | 8 (41) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 5 (6) | 1 (5) | 4 (18) | 6 (10) | 2 (3)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 4 (6) | 7 (8) | 2 (4) | 3 (4) | 5 (13) | 2 (11)
Glossopharyngeal nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (39) | 23 (53) | 5 (11) | 20 (76) | 25 (117) | 6 (21)
Leukoencephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (3) | 0 (0)
Mini mental status examination abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (12) | 2 (2) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (7) | 5 (10) | 3 (6) | 7 (14) | 3 (26) | 1 (1)
Recurrent laryngeal nerve palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus pain (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Taste alteration (Nervous system disorders) | 9 (39) | 12 (67) | 5 (22) | 12 (41) | 10 (70) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (3) | 4 (4) | 2 (6) | 2 (2) | 1 (1) | 2 (2)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 4 (11) | 7 (11) | 2 (4) | 4 (10) | 4 (10) | 0 (0)
Insomnia (Psychiatric disorders) | 6 (27) | 4 (25) | 2 (3) | 9 (31) | 7 (27) | 1 (1)
Bladder hemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (4) | 0 (0)
Bladder pain (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Hemoglobin urine positive (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 0 (0)
Hemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Protein urine positive (Renal and urinary disorders) | 14 (111) | 30 (124) | 17 (67) | 35 (187) | 37 (341) | 12 (70)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urethral pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 5 (12) | 0 (0) | 1 (5) | 5 (5) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Urogenital disorder (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (2) | 3 (10) | 2 (4) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal mucositis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Vaginal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (21) | 1 (2) | 3 (4) | 1 (4) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (31) | 9 (25) | 3 (4) | 6 (14) | 8 (19) | 3 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 10 (18) | 1 (2) | 7 (13) | 9 (12) | 1 (26)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 7 (16) | 19 (76) | 5 (10) | 22 (84) | 21 (83) | 0 (0)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 4 (4) | 1 (1) | 5 (19) | 4 (28) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 5 (6) | 0 (0) | 4 (6) | 2 (3) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 2 (2) | 0 (0) | 3 (3) | 3 (6) | 0 (0)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 (16) | 4 (11) | 1 (1) | 6 (8) | 6 (14) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 3 (50) | 0 (0) | 1 (1) | 3 (4) | 3 (50) | 2 (4)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 5 (21) | 1 (14) | 6 (14) | 4 (5) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (21) | 0 (0) | 1 (1) | 9 (28) | 9 (30) | 2 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (53) | 5 (10) | 0 (0) | 7 (31) | 11 (29) | 0 (0)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (15) | 1 (1) | 2 (7) | 7 (23) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 7 (46) | 7 (42) | 0 (0) | 5 (22) | 7 (89) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (4) | 8 (9) | 1 (2) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (84) | 14 (38) | 4 (13) | 9 (22) | 13 (39) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 9 (90) | 20 (86) | 5 (15) | 21 (86) | 16 (123) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 9 (26) | 15 (42) | 8 (27) | 15 (70) | 25 (122) | 1 (1)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (4) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 2 (3) | 7 (16) | 3 (4) | 6 (11) | 12 (42) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (8) | 1 (1) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (9) | 0 (0) | 1 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (5) | 1 (1) | 0 (0)
Hemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 5 (7) | 2 (2)
Hot flashes (Vascular disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Hypertension (Vascular disorders) | 16 (131) | 34 (174) | 10 (43) | 39 (186) | 35 (365) | 21 (145)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymph leakage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 3 (31) | 3 (13) | 2 (2) | 1 (1) | 3 (14) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-06): https://cdn.clinicaltrials.gov/large-docs/26/NCT01010126/Prot_SAP_000.pdf